CLINICAL TRIAL: NCT01580280
Title: Effect of Upper Cervical and Upper Thoracic Thrust Manipulation Versus Mobilization and Exercise in Patients With Cervicogenic Headache
Brief Title: Manual Therapy and Exercise in Patients With Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Long Island University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/01-006
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic; Headache; Neck Pain; Manipulation; Mobilization; Exercise
MeSH Terms: conditions — Post-Traumatic Headache; Headache; Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thrust manipulation (Experimental)
  Interventions: Other: Thrust Manipulation
- Non-thrust mobilization and exercise (Active Comparator)
  Interventions: Other: Non-thrust Mobilization and Exercise

INTERVENTIONS:
Other: Thrust Manipulation — Upper cervical and upper thoracic thrust manipulation for 6-8 sessions over 2-4 weeks.
  Other Names: High-velocity low-amplitude thrust manipulation of the spine
  Arms: Thrust manipulation
Other: Non-thrust Mobilization and Exercise — Upper cervical and upper thoracic non-thrust mobilization and exercise for 6-8 sessions over 2-4 weeks.
  Other Names: Non-thrust mobilization to cervical and thoracic spines; Cervical range of motion, strength, and postural exercises
  Arms: Non-thrust mobilization and exercise

SUMMARY:
Hypothesis: The group of cervicogenic headache patients receiving upper cervical and upper thoracic thrust manipulation will demonstrate significant and clinically important changes in outcomes when compared to the mobilization and exercise group.

DETAILED DESCRIPTION:
Patients with cervicogenic headache will be randomized to receive 6-8 sessions over 2-4 weeks of either: (1) upper cervical and upper thoracic thrust manipulation, or (2) upper cervical and upper thoracic non-thrust mobilization and range of motion, strength and postural exercises.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervicogenic headache as defined by Cervicogenic Headache International Study Group criteria
* Headache frequency of at least one per week for a minimum of 3 months
* Minimum pain score (NPRS) of 2/10 and minimum disability score (NDI) of 10/50

Exclusion Criteria:

* Bilateral headaches
* Presence of any of the following atherosclerotic risk factors: hypertension, diabetes, heart disease, stroke, transient ischemic attack, peripheral vascular disease, smoking, hypercholesterolemia or hyperlipidemia
* Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e. tumor, fracture, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, etc.)
* History of whiplash injury within the last 6 weeks
* Diagnosis of cervical spinal stenosis
* Bilateral upper extremity symptoms
* Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes)
* Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

  * Muscle weakness involving a major muscle group of the upper extremity.
  * Diminished upper extremity deep tendon reflex of the biceps, brachioradialis, triceps or superficial flexors
  * Diminished or absent sensation to pinprick in any upper extremity dermatome
* Prior surgery to the neck or thoracic spine.
* Involvement in litigation or worker's compensation regarding their neck pain and/or headaches.
* Physical therapy or chiropractic treatment for neck pain or headache in the 3 months before baseline examination.
* Any condition that might contraindicate spinal manipulative therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Headache Frequency | Baseline
  The number of headache days in the past week (as registered in headache diary)
Headache Frequency | 1-week
  The number of headache days in the past week (as registered in headache diary)
Headache Frequency | 4-weeks
  The number of headache days in the past week (as registered in headache diary)
Headache Frequency | 3-months
  The number of headache days in the past week (as registered in headache diary)
Headache Intensity | Baseline
  Average pain intensity as measured by the Numeric Pain Rating Scale (NPRS) per headache episode in the past week.
Headache Intensity | 1-week
  Average pain intensity as measured by the Numeric Pain Rating Scale (NPRS) per headache episode in the past week.
Headache Intensity | 4-weeks
  Average pain intensity as measured by the Numeric Pain Rating Scale (NPRS) per headache episode in the past week.
Headache Intensity | 3-months
  Average pain intensity as measured by the Numeric Pain Rating Scale (NPRS) per headache episode in the past week.
Headache Duration | Baseline
  Average number of headache hours in the last week (as registered in the headache diary)
Headache Duration | 1-week
  Average number of headache hours in the last week (as registered in the headache diary)
Headache Duration | 4-weeks
  Average number of headache hours in the last week (as registered in the headache diary)
Headache Duration | 3-months
  Average number of headache hours in the last week (as registered in the headache diary)
Neck Disability Index (NDI) | Baseline
  Neck pain and disability
Neck Disability Index (NDI) | 1-week
  Neck pain and disability
Neck Disability Index (NDI) | 4-weeks
  Neck pain and disability
Neck Disability Index (NDI) | 3-months
  Neck pain and disability

SECONDARY OUTCOMES:
Global Rating of Change (GROC) | 1-week
  Perceived improvement.
Global Rating of Change (GROC) | 4-weeks
  Perceived improvement.
Global Rating of Change (GROC) | 3-months
  Perceived improvement.
Analgesic Use | Baseline
  Analgesic (medication intake) use per day (as registered in the headache diary).
Analgesic Use | 3-months
  Analgesic (medication intake) use per day (as registered in the headache diary).

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Hagins, PT, PhD, Study Chair — Long Island University
Locations (1):
- Alabama Physical Therapy & Acupuncture, Montgomery, Alabama, United States

REFERENCES:
- [Background] Dunning JR, Cleland JA, Waldrop MA, Arnot CF, Young IA, Turner M, Sigurdsson G. Upper cervical and upper thoracic thrust manipulation versus nonthrust mobilization in patients with mechanical neck pain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):5-18. doi: 10.2519/jospt.2012.3894. Epub 2011 Sep 30. PMID 21979312
- [Derived] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024